CLINICAL TRIAL: NCT06857240
Title: Topical Ruxolitinib Cream for Refractory Cutaneous Dermatomyositis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anthony Fernandez, MD, PhD, Director of Medical Dermatology; W.D. Steck Chair of Clinical Dermatology, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-864
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-07

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Intervention Model Description: Prospective, Single-Arm, Open-Label Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): 1.5 % Ruxolitinib cream
  Interventions: Drug: Ruxolitinib Topical Cream

INTERVENTIONS:
Drug: Ruxolitinib Topical Cream — 1.5% cream

SUMMARY:
This study will assess the safety and efficacy of topical ruxolitinib for treating the refractory cutaneous manifestations in patients with dermatomyositis. The investigators' hypothesis is that topical ruxolitinib will be both safe and effective for such patients.

DETAILED DESCRIPTION:
Dermatomyositis (DM) is an immune-mediated disease that most commonly affects the skin and the muscles. Cutaneous involvement of DM can lead to ulceration with secondary infection, in addition to permanent skin damage in the form of atrophy, scarring, calcinosis, decreased range of motion or lipoatrophy. Furthermore, persistent cutaneous DM is associated with adverse psychological effects and physical symptoms such as pain, burning, and pruritus. The combination of these contribute to a significant negative impact on DM patients' quality of life. Thus, effective treatment of cutaneous DM represents an important therapeutic goal.

Cutaneous DM symptoms and inflammation are often refractory to currently available topical medications . Additionally, continued topical corticosteroid use is associated with well-known adverse effects, including potential worsening of DM-related skin atrophy and adrenal insufficiency.

Recently, topical ruxolitinib has been developed and studied in several dermatologic conditions. In phase 2 and 3 trials in atopic dermatitis, topical ruxolitinib 1.5% cream resulted in significant efficacy in terms of improving both disease activity and itching, without significant side effects. The investigators propose to study use of topical ruxolitinib 1.5% cream as an adjunct for treatment of refractory cutaneous DM lesions in patients who have previously failed other topical medication options.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older with refractory cutaneous symptoms related to either classic dermatomyositis (CD), juvenile dermatomyositis (JD), or amyopathic dermatomyositis (AD). Diagnosis will be based on either Bohan and Peter criteria (CD and JD) or Sontheimer's criteria (AD) (19-22).
* Patients must have had a skin biopsy with histologic features consistent with dermatomyositis and current cutaneous manifestations consistent with dermatomyositis.
* Patients will be considered to have refractory disease if cutaneous manifestations exist despite treatment with systemic corticosteroids and at least one steroid-sparing systemic treatment commonly found to be useful in patients with dermatomyositis. These may include azathioprine, cyclosporine, mycophenolate mofetil, IVIG, methotrexate, hydroxychloroquine, cyclophosphamide, chlorambucil, sirolimus, tacrolimus, and rituximab.
* Patients must have sufficiently active cutaneous involvement of dermatomyositis (BSA>1% to <20%, CDASI activity score > 6, and Physician Global Assessment (PGA) activity score >2).
* Patients must have tried and failed at least one commonly prescribed topical medication in the past, with the last application of a topical medication to active skin lesions occurring greater than 2 weeks prior to enrollment.

  o Commonly prescribed topical medications for dermatomyositis include corticosteroids or calcineurin inhibitors (tacrolimus or pimecrolimus).
* Patients must have been on a stable systemic medication regimen for at least 2 months (60 days) and must agree to keep the regimen stable throughout the study period. As patients with dermatomyositis are commonly treated with combination regimens that include both topical and systemic immunosuppressive medications, any added risk of adverse effects related to ruxolitinib 1.5% cream is considered negligible.
* Patients must be agreeable to use appropriate contraceptive measures while enrolled in the study.

  * Women of childbearing potential must be willing to practice abstinence or use either an oral contraceptive medication or IUD if sexually active.
  * Women of childbearing potential must be willing to have monthly urine pregnancy tests while enrolled in the study
  * Men of childbearing potential must be willing to practice abstinence or use condoms if sexually active.

Exclusion Criteria:

* Patients with dermatomyositis who have minimal-to-no active cutaneous disease (mild involvement with < 1% total body surface area involved and/or CDASI activity score of < 6).
* Patients who have > 20% total BSA involvement of cutaneous dermatomyositis.
* Patients who have used a common prescription topical medication within the previous 2 weeks.
* Patients whose cutaneous findings are not consistent with dermatomyositis and/or have previous biopsy results suggestive of an alternative diagnosis
* Patients not on stable systemic medication regimens for at least 2 months and/or who will not agree to keep the regimen stable throughout the study period.
* Patients who have previously taken a systemic Janus kinase inhibitor but had a poor response, patients who are currently taking systemic Janus kinase inhibitors, or patients who have used a topical Janus kinase inhibitor for their dermatomyositis or any other condition and had poor responses.
* Patients with inflammatory myositis other than dermatomyositis, such as polymyositis or inclusion body myositis.
* Patients with clear features of an overlap autoimmune myositis or with an inflammatory myositis not consistent with dermatomyositis, such as polymyositis or inclusion body myositis.
* Patients with an active malignancy other than non-melanoma skin cancer, or with malignancy-associated dermatomyositis.
* Patients younger than 18 years old

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
CDASI | 8 weeks
  Change in Cutaneous Dermatomyositis Activity and Severity Index (CDASI) activity score (range 0 - 100; higher scores indicate greater disease activity) at 8 weeks

SECONDARY OUTCOMES:
CDASI | week 12
  Change in Cutaneous Dermatomyositis Activity and Severity Index (CDASI) activity score (range 0 - 100; higher scores indicate greater disease activity) at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fernandez, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited IPD will be shared within the publication.
Supporting Information: Study Protocol, SAP
Time Frame: CDSAI-A scores and adverse events at each study assessment point will be included and available in the publication indefinitely.
Access Criteria: Available to all.

REFERENCES:
- [Background] Bailey EE, Fiorentino DF. Amyopathic dermatomyositis: definitions, diagnosis, and management. Curr Rheumatol Rep. 2014 Dec;16(12):465. doi: 10.1007/s11926-014-0465-0. PMID 25366932
- [Background] Robinson ES, Feng R, Okawa J, Werth VP. Improvement in the cutaneous disease activity of patients with dermatomyositis is associated with a better quality of life. Br J Dermatol. 2015 Jan;172(1):169-74. doi: 10.1111/bjd.13167. Epub 2014 Nov 30. PMID 24909747
- [Background] Huber AM, Kim S, Reed AM, Carrasco R, Feldman BM, Hong SD, Kahn P, Rahimi H, Robinson AB, Vehe RK, Weiss JE, Spencer C; Juvenile Dermatomyositis Research Committee of the Childhood Arthritis and Rheumatology Research Alliance. Childhood Arthritis and Rheumatology Research Alliance Consensus Clinical Treatment Plans for Juvenile Dermatomyositis with Persistent Skin Rash. J Rheumatol. 2017 Jan;44(1):110-116. doi: 10.3899/jrheum.160688. Epub 2016 Nov 1. PMID 27803135
- [Background] Sanner H, Sjaastad I, Flato B. Disease activity and prognostic factors in juvenile dermatomyositis: a long-term follow-up study applying the Paediatric Rheumatology International Trials Organization criteria for inactive disease and the myositis disease activity assessment tool. Rheumatology (Oxford). 2014 Sep;53(9):1578-85. doi: 10.1093/rheumatology/keu146. Epub 2014 Mar 31. PMID 24692575
- [Background] Seshadri R, Feldman BM, Ilowite N, Cawkwell G, Pachman LM. The role of aggressive corticosteroid therapy in patients with juvenile dermatomyositis: a propensity score analysis. Arthritis Rheum. 2008 Jul 15;59(7):989-95. doi: 10.1002/art.23829. PMID 18576304
- [Background] Wolstencroft PW, Chung L, Li S, Casciola-Rosen L, Fiorentino DF. Factors Associated With Clinical Remission of Skin Disease in Dermatomyositis. JAMA Dermatol. 2018 Jan 1;154(1):44-51. doi: 10.1001/jamadermatol.2017.3758. PMID 29114741
- [Background] Ladislau L, Suarez-Calvet X, Toquet S, Landon-Cardinal O, Amelin D, Depp M, Rodero MP, Hathazi D, Duffy D, Bondet V, Preusse C, Bienvenu B, Rozenberg F, Roos A, Benjamim CF, Gallardo E, Illa I, Mouly V, Stenzel W, Butler-Browne G, Benveniste O, Allenbach Y. JAK inhibitor improves type I interferon induced damage: proof of concept in dermatomyositis. Brain. 2018 Jun 1;141(6):1609-1621. doi: 10.1093/brain/awy105. PMID 29741608
- [Background] You H, Xu D, Zhao J, Li J, Wang Q, Tian X, Li M, Zeng X. JAK Inhibitors: Prospects in Connective Tissue Diseases. Clin Rev Allergy Immunol. 2020 Dec;59(3):334-351. doi: 10.1007/s12016-020-08786-6. PMID 32222877
- [Background] Hornung T, Janzen V, Heidgen FJ, Wolf D, Bieber T, Wenzel J. Remission of recalcitrant dermatomyositis treated with ruxolitinib. N Engl J Med. 2014 Dec 25;371(26):2537-8. doi: 10.1056/NEJMc1412997. No abstract available. PMID 25539124
- [Background] Kurtzman DJ, Wright NA, Lin J, Femia AN, Merola JF, Patel M, Vleugels RA. Tofacitinib Citrate for Refractory Cutaneous Dermatomyositis: An Alternative Treatment. JAMA Dermatol. 2016 Aug 1;152(8):944-5. doi: 10.1001/jamadermatol.2016.0866. No abstract available. PMID 27120749
- [Background] Paik JJ, Casciola-Rosen L, Shin JY, Albayda J, Tiniakou E, Leung DG, Gutierrez-Alamillo L, Perin J, Florea L, Antonescu C, Leung SG, Purwin G, Koenig A, Christopher-Stine L. Study of Tofacitinib in Refractory Dermatomyositis: An Open-Label Pilot Study of Ten Patients. Arthritis Rheumatol. 2021 May;73(5):858-865. doi: 10.1002/art.41602. Epub 2021 Mar 24. PMID 33258553
- [Background] Dawkins MA, Jorizzo JL, Walker FO, Albertson D, Sinal SH, Hinds A. Dermatomyositis: a dermatology-based case series. J Am Acad Dermatol. 1998 Mar;38(3):397-404. doi: 10.1016/s0190-9622(98)70496-7. PMID 9520020
- [Background] Garcia-Doval I, Cruces M. Topical tacrolimus in cutaneous lesions of dermatomyositis: lack of effect in side-by-side comparison in five patients. Dermatology. 2004;209(3):247-8. doi: 10.1159/000079903. No abstract available. PMID 15459546
- [Background] Barnes L, Kaya G, Rollason V. Topical corticosteroid-induced skin atrophy: a comprehensive review. Drug Saf. 2015 May;38(5):493-509. doi: 10.1007/s40264-015-0287-7. PMID 25862024
- [Background] Hengge UR, Ruzicka T, Schwartz RA, Cork MJ. Adverse effects of topical glucocorticosteroids. J Am Acad Dermatol. 2006 Jan;54(1):1-15; quiz 16-8. doi: 10.1016/j.jaad.2005.01.010. PMID 16384751
- [Background] Kim BS, Howell MD, Sun K, Papp K, Nasir A, Kuligowski ME; INCB 18424-206 Study Investigators. Treatment of atopic dermatitis with ruxolitinib cream (JAK1/JAK2 inhibitor) or triamcinolone cream. J Allergy Clin Immunol. 2020 Feb;145(2):572-582. doi: 10.1016/j.jaci.2019.08.042. Epub 2019 Oct 17. PMID 31629805
- [Background] Kim BS, Sun K, Papp K, Venturanza M, Nasir A, Kuligowski ME. Effects of ruxolitinib cream on pruritus and quality of life in atopic dermatitis: Results from a phase 2, randomized, dose-ranging, vehicle- and active-controlled study. J Am Acad Dermatol. 2020 Jun;82(6):1305-1313. doi: 10.1016/j.jaad.2020.02.009. Epub 2020 Feb 11. PMID 32057960
- [Background] Papp K, Szepietowski JC, Kircik L, Toth D, Eichenfield LF, Leung DYM, Forman SB, Venturanza ME, Sun K, Kuligowski ME, Simpson EL. Efficacy and safety of ruxolitinib cream for the treatment of atopic dermatitis: Results from 2 phase 3, randomized, double-blind studies. J Am Acad Dermatol. 2021 Oct;85(4):863-872. doi: 10.1016/j.jaad.2021.04.085. Epub 2021 May 4. PMID 33957195
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (second of two parts). N Engl J Med. 1975 Feb 20;292(8):403-7. doi: 10.1056/NEJM197502202920807. No abstract available. PMID 1089199
- [Background] Gerami P, Schope JM, McDonald L, Walling HW, Sontheimer RD. A systematic review of adult-onset clinically amyopathic dermatomyositis (dermatomyositis sine myositis): a missing link within the spectrum of the idiopathic inflammatory myopathies. J Am Acad Dermatol. 2006 Apr;54(4):597-613. doi: 10.1016/j.jaad.2005.10.041. Epub 2006 Jan 23. PMID 16546580
- [Background] Euwer RL, Sontheimer RD. Amyopathic dermatomyositis: a review. J Invest Dermatol. 1993 Jan;100(1):124S-127S. doi: 10.1111/1523-1747.ep12356896. PMID 8423381
- [Background] Klein RQ, Bangert CA, Costner M, Connolly MK, Tanikawa A, Okawa J, Rose M, Fakharzadeh SS, Fiorentino D, Lee LA, Sontheimer RD, Taylor L, Troxel AB, Werth VP. Comparison of the reliability and validity of outcome instruments for cutaneous dermatomyositis. Br J Dermatol. 2008 Sep;159(4):887-94. doi: 10.1111/j.1365-2133.2008.08711.x. Epub 2008 Jul 4. PMID 18616782
- [Background] Goreshi R, Okawa J, Rose M, Feng R, Lee LA, Hansen CB, Bangert CA, Connolly MK, Davis MD, Callen JP, Fett NM, Fakharzadeh SS, Clarke JT, Werth VP. Evaluation of reliability, validity, and responsiveness of the CDASI and the CAT-BM. J Invest Dermatol. 2012 Apr;132(4):1117-24. doi: 10.1038/jid.2011.440. Epub 2012 Jan 5. PMID 22217740
- [Background] Carroll CL, Lang W, Snively B, Feldman SR, Callen J, Jorizzo JL. Development and validation of the Dermatomyositis Skin Severity Index. Br J Dermatol. 2008 Feb;158(2):345-50. doi: 10.1111/j.1365-2133.2007.08342.x. Epub 2007 Dec 7. PMID 18067478
- [Background] Rider LG, Werth VP, Huber AM, Alexanderson H, Rao AP, Ruperto N, Herbelin L, Barohn R, Isenberg D, Miller FW. Measures of adult and juvenile dermatomyositis, polymyositis, and inclusion body myositis: Physician and Patient/Parent Global Activity, Manual Muscle Testing (MMT), Health Assessment Questionnaire (HAQ)/Childhood Health Assessment Questionnaire (C-HAQ), Childhood Myositis Assessment Scale (CMAS), Myositis Disease Activity Assessment Tool (MDAAT), Disease Activity Score (DAS), Short Form 36 (SF-36), Child Health Questionnaire (CHQ), physician global damage, Myositis Damage Index (MDI), Quantitative Muscle Testing (QMT), Myositis Functional Index-2 (FI-2), Myositis Activities Profile (MAP), Inclusion Body Myositis Functional Rating Scale (IBMFRS), Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI), Cutaneous Assessment Tool (CAT), Dermatomyositis Skin Severity Index (DSSI), Skindex, and Dermatology Life Quality Index (DLQI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S118-57. doi: 10.1002/acr.20532. No abstract available. PMID 22588740
- [Background] Rider LG, Koziol D, Giannini EH, Jain MS, Smith MR, Whitney-Mahoney K, Feldman BM, Wright SJ, Lindsley CB, Pachman LM, Villalba ML, Lovell DJ, Bowyer SL, Plotz PH, Miller FW, Hicks JE. Validation of manual muscle testing and a subset of eight muscles for adult and juvenile idiopathic inflammatory myopathies. Arthritis Care Res (Hoboken). 2010 Apr;62(4):465-72. doi: 10.1002/acr.20035. PMID 20391500
- [Background] Thomas CL, Finlay AY. The 'handprint' approximates to 1% of the total body surface area whereas the 'palm minus the fingers' does not. Br J Dermatol. 2007 Nov;157(5):1080-1. doi: 10.1111/j.1365-2133.2007.08183.x. Epub 2007 Sep 13. No abstract available. PMID 17854369
- [Background] Yassaee M, Fiorentino D, Okawa J, Taylor L, Coley C, Troxel AB, Werth VP. Modification of the cutaneous dermatomyositis disease area and severity index, an outcome instrument. Br J Dermatol. 2010 Mar;162(3):669-73. doi: 10.1111/j.1365-2133.2009.09521.x. Epub 2009 Oct 26. PMID 19863510

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT06857240/Prot_SAP_000.pdf